CLINICAL TRIAL: NCT00346801
Title: A Phase I Study of Concurrent CPT-11/Cisplatin and Celecoxib With Radiation Therapy for Patients With Unresectable Non-Small Cell Lung Cancer (NSCLC)
Brief Title: CPT-11/Cisplatin and Celecoxib With Radiation Therapy for Patients With Unresectable Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0352
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; Celecoxib; Cisplatin; Platinol; CPT-11; Irinotecan; SC-58635; Celebrex; Radiation Therapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPT-11 + Celecoxib/Cisplatin with RT (Experimental): CPT-11 + Celecoxib + Cisplatin + Radiation Therapy (RT)
  Interventions: Drug: Celecoxib; Drug: Cisplatin; Drug: CPT-11; Radiation: Concurrent Thoracic Radiation Therapy

INTERVENTIONS:
Drug: Celecoxib — 100 mg by mouth (PO) twice daily for 5 days before beginning radiation therapy; continued 7 days per week throughout radiation treatment (about 7 weeks).
  Other Names: Celebrex; SC-58635
Drug: Cisplatin — 25 mg/m^2 IV over 60 minutes on Day 1, Weeks 2-8
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: CPT-11 — 30 mg/m^2 IV over 90 minutes on Day 1, Weeks 2-8, followed by cisplatin which will be infused for 60 minutes.
  Other Names: Irinotecan
Radiation: Concurrent Thoracic Radiation Therapy — 63 Gy at 1.8 Gy/Fx in 35 Fractions over 7 weeks starting 2nd week of celebrex.
  Other Names: XRT; RT

SUMMARY:
Primary Objectives:

* To determine the feasibility, activity, and toxicity of a novel regimen using a concurrent irinotecan (CPT-11)/cisplatin and celecoxib combination for patients with unresectable NSCLC.
* To determine the maximal tolerance dose of celecoxib in patients with unresectable NSCLC treated with irinotecan/cisplatin and concurrent thoracic radiation therapy.
* To correlate the COX-2 expression and other biomarkers with response to the treatment in the tumor from a pretreatment biopsy specimen.

DETAILED DESCRIPTION:
Celecoxib is a non-steroidal-anti-inflammatory drug (NSAIDS), similar to aspirin or ibuprofen. Recent studies have shown that celecoxib has antitumor activity when used alone. It may also increase the tumor sensitivity to radiation, making tumors more responsive to radiation therapy.

Before treatment starts, you will have a complete physical exam, including blood (about 2 teaspoons) and urine tests. You will have a chest x-ray, CT/MRI scans, and/or a PET scan. You may have a bone scan (x-rays of your bones) if your doctor feels it is necessary. You may also have blood tests, x-rays, biopsy of the tumor, and any other tests which your physician feels are necessary for your standard of care.

In this study, you will take celecoxib by mouth for 5 days before beginning radiation therapy. You will continue to receive celecoxib 7 days per week throughout radiation treatment (about 7 weeks). The amount of drug that you take will depend on what dose level you are assigned to. The dose levels are 200mg, 400mg, and 800 mg per day. Ten patients will be treated on each dose level starting at the lower level. You will be required to fill out a medication diary, documenting the dose of celecoxib you are taking and the time that you take it.

You will receive cisplatin and CPT-11 by vein on Day 1 of Weeks 2 through 8. Chemotherapy will be given on an outpatient basis. CPT-11 will be infused by vein over 90 minutes followed by cisplatin which will be infused for 60 minutes. Because cisplatin can cause kidney damage, fluids may need to be injected to "flush" the kidneys. Diuretics are given by vein just before and after receiving cisplatin. So that the physician may better evaluate kidney function during this time, you may be asked to save urine specimens and to keep a record of all fluids taken by mouth during the first 24-48 hours after receiving cisplatin.

Radiation therapy will begin on Day 1 of Week 2 and be given at the same time as chemotherapy. The radiation therapy treatments will be given once a day for 5 days a week, Monday-Friday. The total treatment time for individual patients will be decided by the physician, based on the your general condition and stage of disease. The length of the radiation treatment should be about 7 weeks (35 radiation treatments).

During treatment, you will have blood tests (about 2 teaspoons) every week. You will report to your physician the degree of sore throat, difficulty swallowing, gastric burning, or any symptoms that concern you.

You will be taken off study if the disease becomes worse or side effects become very severe.

After treatment is completed, you will return for follow-up visits at one month, every 3 months for 2 years, every 6 months for 3 to 5 years, then once a year for 10 years. At each follow-up visit, you will have blood (about 2 teaspoons) samples collected for routine lab tests and you will have a chest x-ray. You will have a CT scan of the chest every 6 months. Complete lung function tests will also be done. Lung function tests look at the exchange of the air flow, capacity of the lung, flexibility of the lung, and exchange of oxygen in carbon dioxide in the lungs.

This is an investigational study. All of the drugs in this study are FDA approved and commercially available. The use of these drugs in combination is investigational. Between 30 and 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. No history of active gastric ulcer, active GI bleeding, or renal failure.
2. Patient must have histological or cytological evidence of NSCLC.
3. Nonresectable Stage II or III NSCLC. Inoperable based on patient's physical status is acceptable.
4. KPS is greater than or equal to 70.
5. Age is greater than or equal to 18 or less than or equal to 80.
6. Patient not receiving irradiation therapy or combined modality therapy to treat another malignancy.
7. No evidence of distant metastatic disease.
8. ANC count (segs & bands) is greater than or equal to 2000/mm3 and platelet count is greater than or equal to 100,000/mm3.
9. Serum creatinine less than or equal to 1.5 mg/dL.
10. Total bilirubin is less than or equal to 1.5 times the institutional upper limits of normal value, SGOT less than or equal to 1.5 times the the institutional upper limit of normal.
11. Patients may not be entered on investigational therapeutic trials.
12. Patients or guardian must be informed of and understand the investigational nature of this study and give written informed consent prior to any study procedures.
13. Patient may have prior chemotherapy. Chemotherapy must have been completed 4 weeks prior to study entry.
14. Patients taking cardio-protective dose of aspirin 81 mg are allowed.

Exclusion Criteria:

1. History of poorly controlled hypertension (systolic >150 mm Hg), angina, or other cardiac abnormalities or history of MI or CHF in the last 6 months.
2. General medical or psychological conditions which would not permit the patient to complete the study or sign the informed consent.
3. Pregnancy or women of child bearing potential who do not use an effective (for them) method of birth control throughout their participation in this study.
4. Patients who are currently receiving or have received amifostine for radioprotection within the prior six months are excluded.
5. Patient with history of malignancy other than skin cancer or Carcinoma in-situ within 2 years.
6. Patients who are allergic to Sulfonamides, NSAIDS or Celebrex will be excluded from this protocol.
7. Patients who use routine NSAIDS such as high dose daily use of Aspirin higher than 2 Gm per day will be excluded. Patients will be allowed to take low dose aspirin (less than 200 mg per day).
8. History of cardiovascular diseases that might include one of the following: myocardial infraction, angina, coronary angioplasty, congestive heart failure, stroke, or coronary bypass surgery in the last 6 months.
9. Family history of premature coronary disease (i.e. - onset < 55 years of age).
10. Uncontrolled hypercholesteremia [low-density lipoprotein cholesterol (LDL-C) > 200] more than twice in the repeated tests. Hypercholesteremia needs to be controlled following the updated National Cholesterol Education Program Adult Treatment Panel III Guidelines for at least 3 months prior to enrollment on the study. Hypercholesteremia treatment should continue during the entire period of Celecoxib treatment on the protocol
11. History of deep venous thrombosis, pulmonary embolism, systemic lupus erythematous, family history of protein S or C deficiencies, prior heparin-induced thrombocytopenia, Factor V Leiden deficiencies or high homocysteine levels.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-09; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Celebrex (celecoxib) | 12 week treatment; Continuous assessment and determination of dose-limiting toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Ritsuko R Komaki, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org